CLINICAL TRIAL: NCT05910242
Title: Efficacy and Safety of Remote Ischemic Conditioning in the Treatment of Essential Hypertension
Brief Title: Efficacy and Safety of Remote Ischemic Conditioning in the Treatment of Essential Hypertension (RICBP-EH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RICBP-EH
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC group (Active Comparator): Patients are treated with remote ischemic conditioning (RIC).
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC group (Sham Comparator): Patients are treated with sham remote ischemic conditioning (sham-RIC).
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC group
Procedure: Sham remote ischemic conditioning — Sham-RIC is induced by 4 cycles of 5 min of upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning in the treatment of essential hypertension.

DETAILED DESCRIPTION:
Current studies have shown that remote ischemic conditioning can improve vascular endothelial function, inhibit sympathetic nervous system activity and regulate immune and inflammatory reactions. Thus it may exert anti-hypertensive effects through multiple mechanisms. The purpose of this study is to investigate the efficacy and safety of remote ischemic conditioning on blood pressure patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, regardless of sex;
2. Patients with systolic blood pressure ≥140mmHg with or without taking oral antihypertensive drugs
3. Signed and dated informed consent is obtained

Exclusion Criteria:

1. Secondary hypertension;
2. Clinical blood pressure ≥ 180/110 mmHg or 24-hour mean arterial pressure ≥ 170/100 mmHg;
3. Severe organ dysfunction or failure;
4. Severe hematologic disorders or significant coagulation abnormalities;
5. History of atrial fibrillation or myocardial infarction within 6 months;
6. Individuals who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper limb, acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
7. Individuals who will or have received anticoagulant therapy with drugs such as dabigatran, rivaroxaban, warfarin, etc; ;
8. Pregnant or lactating women;
9. Those who are participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to enrollment;
10. Other conditions that the researchers think are not suitable for the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure | 1-7 days
  Difference in mean systolic blood pressure during RIC/sham-RIC between two groups.

SECONDARY OUTCOMES:
Mean diastolic blood pressure | 1-7 days
  Difference in mean diastolic blood pressure during RIC/sham-RIC between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Yin WJ, Wang SJ, Qu Y, Ren JX, Zhang P, Abuduxukuer R, Yang Y, Guo ZN. Efficacy of remote ischemic conditioning on blood pressure in essential hypertension in China (RICBP-EH): a randomised, controlled, parallel-group trial. EClinicalMedicine. 2025 Oct 16;89:103562. doi: 10.1016/j.eclinm.2025.103562. eCollection 2025 Nov. PMID 41146928